CLINICAL TRIAL: NCT02410304
Title: Pragmatic Study Comparing the Clinical Evlauation Methods ( C) and / or Ultrasound Method ( B or D) in Rheumatoid Arthritis (RA) to Adapt Treatment
Brief Title: Pragmatic Study Comparing the Clinical Evlauation Methods ( C) and / or Ultrasound Method ( B or D) in Rheumatoid Arthritis to Adapt Treatment
Acronym: BCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BCD 29BRC14.0097
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis / ultrasonography / synovitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis | interventions — Diagnostic Imaging; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm C (Clinical) (Other): No drug and no placebo were used in this arm. Patients were followed only by clinical évaluation.
  Interventions: Device: Xrays
- Arm B (Clinical + Ultrasound) (Other): No drug and no placebo were used in this arm. Patients were followed by Clinical evaluation in combination with ultrasound (in B mode).
  Interventions: Device: Xrays; Device: Ultrasound (B mode )
- Arm D (Ultrasound) (Other): No drug and no placebo were used in this arm. Patients were followed by Ultrasound approach in D mode.
  Interventions: Device: Ultrasound (D mode)

INTERVENTIONS:
Device: Xrays — Clinical evaluation
  Arms: Arm B (Clinical + Ultrasound); Arm C (Clinical)
Device: Ultrasound (B mode )
  Arms: Arm B (Clinical + Ultrasound)
Device: Ultrasound (D mode)
  Arms: Arm D (Ultrasound)

SUMMARY:
This study compares different methods of clinical evaluation (C) and/or ultrasound (B or D) concerning the rheumatoid arthritis in order to monitore the treatment. This study will provide the exact number of patients in remission according the 3 methods.

It could allow to assess the concordance between the 3 evaluated methods. This study will permit to define the best method which limit the evolution of structural damages ( principal criteria).

DETAILED DESCRIPTION:
The aim of this study is to evaluate the Xrays evolution at 1 year ( at least one new erosion versus no erosion with the Sharp modified by van der Heijde) of patients affected by rheumatoid arthritis (ACR/EULAR 2010). The first approach is the assessment of remission defined by modified SDAI in order to evaluate in all cases the same number of joints [Simplified Disease Activity Index algebric sum of 5 parametres : number of painful joints (28 joints) , number of synovitis (38 joints), global evaluation of patient and and practitioner with VAS, and PCR ≤ 3.3mg/l] (mode C). The second one is a combined approach: clinical-ultrasound (same criteria but with MTPs and shoulders in B mode so a 26 joints evaluation with clinical examination and 12 joints evaluation in B mode) (mode B). The last one is an ultrasound approach (remission defined as the absence of power Doppler on 38 joints (28 of SDAI plus 10 MTPs joints) (mode D) in a pragmatical context (study assessed by private rheumatologists and hospital rheumatologists).

This trial is a National randomized multicentre trial that compares three modes of follow to adjust the therapeutic adaptation in Rheumatoid Artritis.

ELIGIBILITY:
* Inclusion Criteria:

  * Both gender patients aged 18 -to 80 years old
  * Patients will be eligible if they fulfill ACR/EULAR 2010 rheumatoid arthritis
  * All the treatment recommended for rheumatoïd arthritis (anti-inflammatory drugs, steroids, hydroxychloroquine, salazopyrine, methotrexate, ARAVA or biologics treatment: Enbrel, humira, remicade, cimzia, tocilizumab, rituximab, abatacept, simponi) would be in stable posology since at least 12 weeks before inclusion
  * Patients would be able to understand and be agree with the protocole
  * Patients would be able to consent
* Exclusion Criteria:

  * Patient unable to cooperate patient and who refuse to sign consent form
  * Patient unable to understand the study,under administrative supervision or legal guardianship
  * Signs and symptoms of uncontroled or severe progressive pathology at the level of renal, hepatic, hematological, endocrine, lung, cardiac, neurological or cerebral
  * Scheduled surgery procedure during the study on the estimated joint.
  * Patient non-affiliated to social security
  * Pregnant and nursing mothers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2015-10-06 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Assessement of the Xrays evolution at 1 year through adaptated treatment according to clinical or ultrasound remission criteria. | 1 year
  The primary outcome is to evaluate the Xrays evolution at 1 year ( at least one new erosion versus no erosion with the Sharp modified by van der Heijde) of rheumatoid arthritis patients (ACR/EULAR 2010) according to remission defined by modified SDAI in order to evaluate in all cases the same number of joints [Simplified Disease Activity Index algebric sum of 5 parametres : number of painful joints (28 joints) , number of synovitis (38 joints), global evaluation of patient and practitioner with VAS, and PCR ≤ 3.3mg/l] (mode C), with a combined approach clinical-ultrasound (same criteria but with MTPs and shoulders in B mode so a 26 joints evaluation with clinical examination and 12 joints evaluation in B mode) (mode B) or an ultrasound approach (remission défined as the absence of power Doppler on 38 joints (28 of SDAI plus 10 MTPs joints) (mode D) in a pragmatical context (study assessed by private rheumatologists and hospital rheumatologists).

SECONDARY OUTCOMES:
Evaluation of the proportion of rheumatoid arthristis in remission according to the method used | at 3 month, 6 month, 9 month and 1 year
Assessement of the Xrays evolution at 2 years | 2 years

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Angers, Angers
  - CHRU Brest, Brest
  - CHU La Roche sur Yon, La Roche-sur-Yon
  - CH Le Mans, Le Mans
  - CH de Lorient, Lorient
  - CHU Nantes, Nantes
  - CHR Orléans, Orléans
  - CHU SUD Rennes, Rennes
  - CHU Tours, Tours
  - CH Vannes, Vannes